CLINICAL TRIAL: NCT05953610
Title: Endotypic Traits and Obstructive Sleep Apnea Surgery
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Eric J. Kezirian, MD, MPH, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1.0; R01HL160993 (NIH)
Record Dates: First submitted 2023-05-08; First posted 2023-07-20 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Obstructive Sleep Apnea
Keywords: surgery; loop gain; arousal threshold
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Acetazolamide; Eszopiclone

STUDY DESIGN:
Intervention Model Description: Prospective cohort study will include an anticipated 150 study participants undergoing soft palate surgery. The randomized crossover (interventional) study will include the anticipated 90 who do not achieve successful treatment of their obstructive sleep apnea with surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acetazolamide (Experimental): Treatment with acetazolamide 500 mg nightly for 1 month.
  Interventions: Drug: Acetazolamide 500 MG QHS
- Acetazolamide/Eszopiclone (Experimental): Treatment with acetazolamide 500 mg and eszopiclone 3 mg nightly for 1 month.
  Interventions: Drug: Acetazolamide 500 MG QHS; Drug: Eszopiclone 3 mg QHS

INTERVENTIONS:
Drug: Acetazolamide 500 MG QHS — Acetazolamide
Drug: Eszopiclone 3 mg QHS — Eszopiclone
  Arms: Acetazolamide/Eszopiclone

SUMMARY:
This study will examine factors associated with outcomes after soft palate surgery and medications (acetazolamide, eszopiclone) that may treat other potential causes of obstructive sleep apnea (loop gain, arousal threshold).

DETAILED DESCRIPTION:
This is a prospective cohort (observational) study of 150 participants with moderate to severe obstructive sleep apnea (OSA) unable to tolerate positive airway pressure who are undergoing drug-induced sleep endoscopy (DISE), including measurement of upper airway closing pressure (Pclose), and tissue-repositioning soft palate surgery. Before and 6 months after surgery, the investigators will measure OSA severity (apnea-hypopnea index) with sleep studies (polysomnograms). Using a recently-validated polysomnography-based signal processing algorithm, the investigators will systematically assess the underlying mechanisms of OSA (traits) and airflow shape (consistent with palate obstruction). The expected 90 participants without resolution of OSA after surgery (surgery failures) will participate in an experimental randomized crossover study of acetazolamide (1 month) and acetazolamide/eszopiclone combination (1 month). Polysomnograms will be performed with each treatment, with algorithm-based determination of traits.

ELIGIBILITY:
Inclusion criteria are:

1. age ≥21 years;
2. moderate to severe OSA (obstructive AHI ≥ 15 events/hour);
3. central/mixed apnea index <5 events/hour;
4. intolerance of positive airway pressure (defined as use < 2 hours/night at least 5 nights/week);
5. intolerance or poor candidate for oral appliance;
6. participant has provided informed consent for palate surgery as part of their standard of care;
7. tonsil size 0-2+ (without markedly enlarged tonsils that have high surgical success rates);
8. DISE without evidence of complete tongue-related obstruction (reflecting poorer results with isolated palate surgery);
9. medications stable for ≥2 months;
10. body mass index <35 kg/m2;
11. absence of uncontrolled nasal obstruction;
12. no prior pharyngeal surgery other than tonsillectomy;
13. no neurologic, cardiac or pulmonary disorders;
14. absence of psychiatric disorder except for treated depression or mild anxiety;
15. no co-existing sleep disorder, such as narcolepsy, chronic insomnia, or restless legs syndrome;
16. no use of hypnotics, anxiolytics, stimulants, or sedating antidepressants;
17. no near-miss or prior motor vehicle crash due to sleepiness in past 12 months; and
18. <3 caffeinated beverages daily.

Exclusion criteria are:

1. history of allergic reaction to either of the study drugs;
2. subjects with prior serious allergic reaction (such as Stevens-Johnson syndrome) to sulfonamides;
3. subjects with a history of hypersensitivity to either of the two study drugs;
4. subjects who are on high-dose aspirin therapy due to risk of severe metabolic acidosis;
5. subjects with severe kidney disease or severe liver disease;
6. subjects with a history of electrolyte imbalance or adrenal insufficiency (due to risks related to acetazolamide);
7. subjects on ketoconazole or other strong CYP3A4 inhibitors (these will increase eszopiclone blood levels);
8. pregnancy; and
9. alcohol or substance abuse.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-01-07 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Apnea-hypopnea index | 6 months
  apneas plus hypopneas per hour of sleep

OTHER OUTCOMES:
Pclose | 6 months
  upper airway closing pressure, as measured with administration of positive airway pressure therapy and observation of airway dimensions with flexible fiberoptic endoscopy
Vpassive | 6 months
  ventilation at normal ventilatory drive, as measured using software to analyze raw polysomnogram data
Loop gain | 6 months
  ventilatory drive response to a 1 cycle/min reduction in ventilation (ventilatory control), as measured using software to analyze raw polysomnogram data
Arousal threshold | 6 months
  median ventilatory drive immediately preceding scored EEG arousals (propensity to wake up), as measured using software to analyze raw polysomnogram data

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - UCLA Santa Monica Medical Center, Santa Monica, California
  - UCLA Westwood, Westwood, Los Angeles, California